CLINICAL TRIAL: NCT01867853
Title: Volume Responsiveness Before Spontaneous Breath Trial Predicts the Outcome of Mechanical Ventilation Weaning in Critically Ill Patients
Brief Title: Volume Responsiveness Before SBT Predicts the Outcome of Mechanical Ventilation Weaning in Critically Ill Patients
Acronym: weaning
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Collaborators: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Director, Southeast University, China
Other Study IDs: 10286
Record Dates: First submitted 2013-05-06; First posted 2013-06-04 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Weaning Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- successful weaning: the SUCCESS of SBT or not need for reintubation or noninvasive ventilation within 48 h following extubation
  Interventions: Device: PLR
- failed weaning: the failure of SBT or the need for reintubation or noninvasive ventilation within 48 h following extubation
  Interventions: Device: PLR

INTERVENTIONS:
Device: PLR — passive leg raising test was done before and at the end of SBT
  Other Names: passive leg raising

SUMMARY:
To evaluate the performance of volume responsiveness in predicting the outcome of mechanical ventilation weaning in critically ill patients.

DETAILED DESCRIPTION:
82 patients, 61 succeed and 21 failed

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilation

Exclusion Criteria:

* pregnancy or breast-feeding
* tracheostomy at baseline
* myasthenia gravis or acute polyradiculoneuropathy
* end-stage chronic illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients were mechanically ventilated and ready to undergo a spontaneous breathing trial (SBT) with a T-piece
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
changes of cardiac index | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin DOU, Principal Investigator — Southeast University
Locations (1):
- Zhongda hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Result] MacIntyre N. Discontinuing mechanical ventilatory support. Chest. 2007 Sep;132(3):1049-56. doi: 10.1378/chest.06-2862. PMID 17873200
- [Result] Eskandar N, Apostolakos MJ. Weaning from mechanical ventilation. Crit Care Clin. 2007 Apr;23(2):263-74, x. doi: 10.1016/j.ccc.2006.12.002. PMID 17368170
- [Result] MacIntyre NR, Cook DJ, Ely EW Jr, Epstein SK, Fink JB, Heffner JE, Hess D, Hubmayer RD, Scheinhorn DJ; American College of Chest Physicians; American Association for Respiratory Care; American College of Critical Care Medicine. Evidence-based guidelines for weaning and discontinuing ventilatory support: a collective task force facilitated by the American College of Chest Physicians; the American Association for Respiratory Care; and the American College of Critical Care Medicine. Chest. 2001 Dec;120(6 Suppl):375S-95S. doi: 10.1378/chest.120.6_suppl.375s. No abstract available. PMID 11742959
- [Result] Monnet X, Teboul JL, Richard C. Cardiopulmonary interactions in patients with heart failure. Curr Opin Crit Care. 2007 Feb;13(1):6-11. doi: 10.1097/MCC.0b013e328013c865. PMID 17198043
- [Result] Teboul JL, Monnet X. Detecting volume responsiveness and unresponsiveness in intensive care unit patients: two different problems, only one solution. Crit Care. 2009;13(4):175. doi: 10.1186/cc7979. Epub 2009 Aug 10. PMID 19678915
- [Result] Monnet X, Teboul JL. Passive leg raising. Intensive Care Med. 2008 Apr;34(4):659-63. doi: 10.1007/s00134-008-0994-y. Epub 2008 Jan 23. PMID 18214429